CLINICAL TRIAL: NCT03275883
Title: Retrospective Analysis to Identify Independent Predictive Risk Factors for Early and Late Arterial Occlusion in Liver Transplantation and Compare Short and Long-term Outcomes for Aorto-hepatic Conduits in Liver Transplantation
Brief Title: Arterial Patency in Liver Transplantation
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: University Hospital Birmingham NHS Foundation Trust (Other); Medical University Innsbruck (Other); University of Bologna (Other); The Leeds Teaching Hospitals NHS Trust (Other); University of California, Los Angeles (Other); Johannes Gutenberg University Mainz (Other); Rennes University Hospital (Other); University of Lyon (Other); University of Rochester (Other); University of Southern California (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-01889
Record Dates: First submitted 2017-09-05; First posted 2017-09-08 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Aortohepatic Conduit; Patency Rate; Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Aortohepatic Conduit — Placement of an interposition graft between hepatic artery and aorta during liver transplantation

SUMMARY:
The aim of this study is to determine the risk profile of hepatic artery occlusion in liver transplant recipients who received an aortohepatic conduits, analyzing all consecutive cadaveric liver transplantations from July 2007 to 31st December 2016. Medical records will be examined and adverse events will be analyzed and categorized using the Clavien-Dindo classification and Comprehensive Complication Index.

DETAILED DESCRIPTION:
BACKGROUND

Arterial conduits in liver transplantation are almost as old as the procedure itself. First described by Starzl in 1984, the knowledge remains superficial. Although rarely performed, there is no doubt that thousands of patients' lives were saved because of the use of arterial grafts. However, arterial grafts are known to be associated with a higher rate of occlusion and a lower patient and graft survival when compared to conventional end-to-end anastomosis. In our recent retrospective study, the investigators showed that retransplantation procedure and aspirin in patients' medication are independent risk factors for the need of an arterial conduit. The investigators assume that aspirin could be a surrogate marker for vascular and metabolic status. Furthermore, in a meta-analysis the investigators found a four times higher occlusion rate compared to non-conduits.

Whether the site of conduit placement or certain types of material have an impact on occlusion and graft survival remains unknown. In addition, several studies discuss that antiaggregation or anticoagulation might be protective for occlusion of arterial conduits. Currently, there is no study that investigated this problem, most probably because of low case numbers.

STUDY OBJECTIVES

The primary goal of this study is to conduct a multicenter cohort analysis to define the outcome of different types of conduits and to investigate whether antiplatelet / anticoagulantion has an impact on patency rates.

1. Specific aim #1: To identify independent risk factors for early and late occlusion of arterial conduits in liver transplantation.
2. Specific aim #2: To compare different placement sites (infrarenal, supraceliac, iliacal, etc.) of arterial conduits in terms of occlusion rates and graft survival.
3. Specific aim #3: To investigate whether antiplatelet therapy is protective in terms of arterial patency.

STUDY DESIGN

This will be a multicenter single cohort study including only cases of deceased donor liver transplantation that required an aorto-hepatic or iliac-hepatic conduit for arterial reconstruction. Primary endpoint is 30-day conduit patency. Secondary endpoints include postoperative complications, death, late conduit occlusion, graft and patient survival.

SETTING

This multicenter cohort study will include several high-volume centers worldwide. Each participating center requires a prospective database from that data can be extracted. All consecutive cases of deceased donor liver transplantation requiring an arterial conduit from 1st of January 2007 until 31st of December 2016 are included allowing a minimum follow-up time of 6 months. Data collection at conduit4olt.org will be prospective, structured, anonymized, and encrypted.

INSTITUTIONAL REVIEW POLICY / ETHICAL POLICY

Each participating center is responsible to contact their local ethics committee and receive approval for participation, if applicable. For example, this project is considered as an audit in some countries and thus there is no need for formal approval in the form of a protocol submission.

ELIGIBILITY CRITERIA

Inclusion criteria:

* Liver transplantation requiring aorto-hepatic or iliac-hepatic conduits
* Deceased donor after brain death (DBD) or deceased donor after circulatory death (DCD)
* Whole organ as well as split allografts
* Primary liver transplantation as well as liver retransplantation
* Recipient age ≥18 years

Exclusion criteria:

* Living donor liver transplantation
* Pediatric liver transplantation (recipient age <18 years)
* Arterial reconstruction other than aorto-hepatic or iliac-hepatic conduits
* Multivisceral transplantations

ESTIMATED SAMPLE SIZE

Each center should provide at least 30 cases that meet the inclusion criteria to allow adequate event rates for each outcome.

Statistical methods

The primary and secondary endpoints will be compared with patient and operation characteristics with univariate analysis. ROC Curve analysis will be performed to dichotomize continuous variables. Multivariable analysis (binary logistic and Cox regression) will be performed to identify independent risk factors. Statistical analysis will be performed using R Studio version 1.0.44 (RStudio, Inc. GNU Affero General Public License v3, Boston, MA, 2016) with the graphical user interface rBiostatistics.com beta version (rBiostatistics.com, Zurich, Switzerland, 2016, GNU License).

Christian E. Oberkofler Tim Reese Dimitri A. Raptis Henrik Petrowsky

On behalf of the conduit4olt.org team Swiss HPB Center, Department of Surgery and Transplantation, University Hospital Zurich, Switzerland

ELIGIBILITY:
Inclusion Criteria:

* Liver transplantation requiring aorto-hepatic or iliac-hepatic conduits
* Deceased donor after brain death (DBD) or deceased donor after circulatory death (DCD)
* Whole organ as well as split allografts
* Primary liver transplantation as well as liver retransplantation
* Recipient age ≥18 years

Exclusion Criteria:

* Living donor liver transplantation
* Pediatric liver transplantation (recipient age <18 years)
* Arterial reconstruction other than aorto-hepatic or iliac-hepatic conduits
* Multivisceral transplantations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who recieved an aorto-hepatic conduit during liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 567 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Independent risk factors | June 2007 til 31st December 2016
  To identify independent risk factors for early and late occlusion of arterial conduits in liver transplantation.
Placement sites | June 2007 til 31st December 2016
  To compare different placement sites (infrarenal, supraceliac, iliacal, etc.) of arterial conduits in terms of occlusion rates and graft survival
Patency Rates | June 2007 til 31st December 2016
  To investigate whether antiplatelet therapy is protective in terms of arterial patency.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
URL: http://conduit4olt.org